## Reinfection rates of soil-transmitted helminth infections among school aged-children following a single or a 4-monthly health hygiene education: an open label clinical trial



## Participant Information Sheet and Informed Consent

Inke Nadia D. Lubis, MD, PhD
Rizky Keumala Ansari Nasution, MD
Badai Buana Nasution, MD
Hendri Wijaya, MD
Aridamuriany D. Lubis, MD
Munar Lubis, MD

Universitas Sumatera Utara Medan, Indonesia 2019 **Participant Information Sheet** 

Sir/Madam,

My name is Dr. Rizky Keumala Ansari Nasution from Department of Paediatrics, Faculty of Medicine, Universitas Sumatera Utara, Medan, Indonesia. We are currently run a study entitled "Reinfection rates of soil-transmitted helminth infections among school-aged children following a single or a 4-monthly health hygiene education: an open label clinical trial".

Soil-transmitted helminth (STH) infections remain high among children. Indonesia is one of the countries with high prevalence rates. Helminth infection affect the growth, concentration, intellectual and child participation in school. Therefore your child is being invited to take part in a research study. We will assess whether your child is infected with STH using an examination from the stool by looking the STH eggs in the stool using microscopy. If we found your child is infected with helminth, we will treat your child accordingly. We will also give education to your child so we can prevent further STH infection.

In this study, all information about your child will be kept strictly confidential. All expenses for the examination and treatment will be free of charge. You have the right to refuse consent in the study.

If you agree to participate, we ask you to sign the informed consent.

Study investigator

Dr. Rizky Keumala Ansari Nasution

## **Informed Consent**

Study title: Reinfection rates of soil-transmitted helminth infections among school-aged children following a single or a 4-monthly health hygiene education: an open label clinical trial

I give consent to the above study:

| Name<br>Age / Sex<br>Address | :<br>:<br>: | years, Male / Female |
|---|---|---|
| To my child:<br>Name<br>Age / Sex<br>Address | :<br>: | years, Male / Female |
| I confirm that the I have read and understand the participant information sheet and that the participation is voluntary. | | |
| | o volumaly. | |
| | | ,2019 |
| Name of study investig | gator | Name of parent/guardian |
| Signature | | Signature |
| dr. Rizky Keumala Ansari | Nasution | |